CLINICAL TRIAL: NCT03286283
Title: A Prospective, Multicenter, Single Arm Clinical Study Evaluating the Use of J-Plasma® for Dermal Resurfacing
Brief Title: The Use of J-Plasma® for Dermal Resurfacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apyx Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-1558
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Results first posted 2019-08-07 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Facial Wrinkles; Rhytides
Keywords: Rhytides; Wrinkle Reduction; J-Plasma; Dermal Resurfacing

STUDY DESIGN:
Intervention Model Description: This is a multi-center, single arm, evaluator-blind prospective study of 55 study subjects who are seeking a procedure to reduce the appearance of wrinkles and rhytides. Enrolled study subjects will receive one procedure with J-Plasma at enrollment. Wrinkle severity will be assessed using the Fitzpatrick Wrinkle and Elastosis Scale (FWS) at baseline and at each follow-up time point. Scores at each follow-up time point will be compared to the scores at baseline for each enrolled subject.
Masking Description: This is a single-arm study in which investigators are not blinded. However, blinded Independent Photographic Reviewers (IPR) will be utilized to review all images (baseline and all follow-up time points) and assign FWS scores.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- J-Plasma (Experimental): Each study subject will receive one procedure with J-Plasma at enrollment.
  Interventions: Device: J-Plasma

INTERVENTIONS:
Device: J-Plasma — Dermal resurfacing procedure with J-Plasma.
  Other Names: Cold Helium Plasma

SUMMARY:
This study evaluates the safety and effectiveness of J-Plasma in the reduction of facial wrinkles and rhytides. It is a multi-center, single arm, evaluator-blind prospective study of 55 study subjects who are seeking a procedure to reduce the appearance of wrinkles and rhytides and will be conducted at up to 5 investigational centers in the United States. Each study subject will receive one procedure with J-Plasma at enrollment. Follow-up will occur immediately following the procedure, at 10 days, 1, 3, and 6 months after enrollment.

DETAILED DESCRIPTION:
The study objective is to demonstrate the safety and efficacy of the J-Plasma system for use in dermal skin resurfacing.

This is a multi-center, single arm, evaluator-blind prospective study of 55 study subjects who are seeking a procedure to reduce the appearance of wrinkles and rhytides at up to 5 investigational centers in the United States.

Study subjects that meet study eligibility criteria and have provided informed consent will be enrolled in the study. During the procedure, the investigators will use J-Plasma on applicable facial zones to reduce wrinkles and rhytides.

Study subjects will be followed immediately following the procedure, at 10 days, 1, 3, and 6 months post-procedure for study assessments.

Study enrollment is expected to occur over 3-6 months. Imaging and study assessments will continue through 6 months post-procedure. Total study duration is expected to be approximately 9-12 months.

Primary study endpoints will be assessed at 3 months following the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥30 years of age.
2. Subject is seeking improvement of facial appearance by reducing facial wrinkles and rhytides.
3. Subject with a facial wrinkle score rating of at least 2 on the FWS as determined by the investigator.
4. Subject with a Fitzpatrick Skin Scale score ≤III.
5. Subject is willing and able to provide written informed consent.
6. Subject is willing and able to comply with protocol requirements, including obtaining study-required images/photos and assessments, and returning for follow-up visits.
7. Subject is willing to release rights to study Sponsor for the use of the photos, including in potential publication.
8. Subject is willing to abstain from other facial cosmetic procedures through the 6 month follow-up visit; examples include, but are not limited to, laser or chemical re-surfacing, dermabrasion, neuromodulator and/or filler injections, aesthetic facial surgery, etc.

Exclusion Criteria:

1. Subject with a Fitzpatrick Skin Scale score >III.
2. Subject is pregnant or lactating.
3. Active HSV-1 or diabetes mellitus.
4. Active cut, wound, or infection on the skin of the face.
5. Subject has used, within the past 30 days, Accutane or any medication that can cause dermal hypersensitivity.
6. Subject has a history of autoimmune disease.
7. Subject with a bleeding disorder or who is on blood thinning medication that may be at risk for bleeding.
8. Subject has a known adverse reaction to anesthetics.
9. Subjects with active skin disease of the facial area or known connective tissue disease.
10. Subjects with known susceptibility to keloid formation or hypertrophic scarring.
11. Subjects with present cancerous or pre-cancerous lesions in the area to be treated.
12. Subject who, for any reason, suspects that they will not be able to complete the prescribed follow-up assessment(s);
13. Subject has had concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety and efficacy of the study treatment method.
14. Subject is not willing to release rights to study Sponsor for the use of the photos, including in potential publication.
15. Subject is enrolled in another investigational (drug or device) clinical trial that can interfere with this study's assessments.
16. Subject has undergone a facelift procedure or received facial injections within the past year.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Ponce, BS(ACS), Study Director — Apyx Medical (formerly Bovie Medical Corporation)
Locations (3):
- United States (3):
  - Miami Plastic Surgery, Miami, Florida
  - Institute for Integrated Aesthetics, Sarasota, Florida
  - Atlanta Dermatology, Vein & Research Center, Alpharetta, Georgia

IPD SHARING:
Plan to Share IPD: No
The Sponsor does not plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Holcomb JD, Kelly M, Hamilton TK, DeLozier JB 3rd. A Prospective Study Evaluating the Use of Helium Plasma for Dermal Resurfacing. Lasers Surg Med. 2020 Dec;52(10):940-951. doi: 10.1002/lsm.23257. Epub 2020 Apr 29. PMID 32350901

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who were enrolled were assigned to a/the treatment group.
Period: Overall Study
Arm/Group | J-Plasma
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- J-Plasma: Each study subject received one procedure with J-Plasma at enrollment.
  J-Plasma: Dermal resurfacing procedure with J-Plasma.
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants] — Adults 30 years of age or older who provided informed consent and who met the inclusion/exclusion criteria.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 37
    >=65 years | 18
Age, Continuous [Mean (Full Range); unit: years] | 61.5 [31 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity are not mutually exclusive categories.
  Participants
    American Indian/Alaskan Native | 1
    Hispanic or Latino | 10
    White | 48
Region of Enrollment [Number; unit: participants]
  United States | 55
Fitzpatrick Wrinkle and Elastosis Scale (FWS) Score [Count of Participants; unit: Participants] — Participants' Average Fitzpatrick Wrinkle and Elastosis Scale (FWS) score at baseline as determined by Independent Photographic Reviewers; the FWS is a scale of 1 to 9 where 9 represents the highest severity of wrinkles and rhytides and 1 represents the lowest severity of wrinkles and rhytides.
  Participants
    Baseline FWS Score = 1 | 1
    Baseline FWS Score = 2 | 2
    Baseline FWS Score = 3 | 1
    Baseline FWS Score = 4 | 10
    Baseline FWS Score = 5 | 4
    Baseline FWS Score = 6 | 1
    Baseline FWS Score = 7 | 8
    Baseline FWS Score = 8 | 20
    Baseline FWS Score = 9 | 8

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Fitzpatrick Wrinkle and Elastosis Scale (FWS) Score
Description: The comparison of the proportion of subjects (i.e. percentage of treatment responders) with a ≥ 1-score improvement on the FWS at the 3-month visit, as compared to baseline as determined by at least 2 out of 3 blinded Independent Photographic Reviewers. Min=1, Max=9, where 1 is best and 9 is worst. The larger the difference between the baseline and 3 month scores, the greater the improvement.
Time Frame: Baseline to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
Participants | 51

2. Primary Outcome: Adverse Event Rate and Duration
Description: Adverse event rates, categorized by duration
Time Frame: Up to 3 months
Measure: Number; unit: percentage of adverse events
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
percentage of adverse events
  Percentage of Serious Adverse Events | 0
  Percentage of Adverse Events Resolved in 7 Days | 41.8
  Percentage Adverse Events Resolved in 14 Days | 58

3. Secondary Outcome: Number of Participants With a ≥ 1-score Improvement on the Fitzpatrick Wrinkle and Elastosis Scale (FWS) and at Least an "Improved" Rating on the Modified Global Aesthetic Improvement Scale (GAIS) at the 3-month Visit.
Description: Assessment of modified Global Aesthetic Improvement Scale (GAIS) at the 3-month visit compared to baseline as assessed by the investigator. Scale ratings: "Very much improved," "Much improved," "Improved," "No change," "Worse," "Much worse," and "Very much worse." An "improvement" on the modified GAIS includes "Improved," "Much improved," or "Very much improved."
Time Frame: Baseline to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
Participants | 53

4. Secondary Outcome: Evaluation of Pain and Discomfort
Description: The evaluation of the pain and discomfort after treatment as reported by the subject on a 10-point visual analog scale (VAS). Mean change in VAS from baseline to 3 months. 0 = best possible level of pain and discomfort, 10= worst possible level of pain and discomfort.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
score on a scale | -3.8 (3.0)

5. Other Pre Specified Outcome: Number of Participants With an Improvement on the FWS (as Scored by Independent Reviewers) and Modified GAIS Scale (as Scored by Participants) at 3 Months
Description: Fitzpatrick Wrinkle and Elastosis Scale (FWS) ≥ 1-score improvement and ≥ 75% agreement with at least an "improved" rating by the subject on the modified Global Aesthetic Improvement Scale (GAIS) at 3 months compared to baseline. FWS Scale: Min=1, Max=9, where 1 is best and 9 is worst. The larger the difference between the baseline and 3 month scores, the greater the improvement. Modified GAIS Scale ratings: "Very much improved," "Much improved," "Improved," "No change," "Worse," "Much worse," and "Very much worse." An "improvement" on the modified GAIS includes "Improved," "Much improved," or "Very much improved."
Time Frame: Baseline to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
Participants | 50

6. Other Pre Specified Outcome: Mean Change in Fitzpatrick Wrinkle and Elastosis Scale (FWS) From Baseline to 3-month Follow-up Visit
Description: Magnitude of improvement measured by the mean change in Fitzpatrick Wrinkle and Elastosis Scale (FWS) from baseline to 3-month visit. Scale of 1 to 9 where 1 represents the lowest severity of wrinkles and 9 represents the greatest severity of wrinkles. Negative change value represents aesthetic improvement.
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
units on a scale | -2.13 (1.02)

7. Other Pre Specified Outcome: Study Subject Satisfaction at 3-month Visit
Description: Evaluation of the subject satisfaction as reported by the subject on a visual analog scale (VAS). VAS scale ranges 0-10, 0 = best possible level of satisfaction, 10= worst possible level of satisfaction
Time Frame: 3 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
score on a scale | 2.5 (3.0)

8. Other Pre Specified Outcome: Achievement of Re-epithelialization - 10 Days
Description: Achievement of re-epithelialization by facial zone and across facial zones after treatment
Time Frame: 10 Days
Measure: Mean (Standard Deviation); unit: percentage of re-epithelialization
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
percentage of re-epithelialization | 96.8 (5.7)

9. Other Pre Specified Outcome: Achievement of Re-epithelialization - 1 Month
Description: Achievement of re-epithelialization by facial zone and across facial zones after treatment
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: percentage of re-epithelialization
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
percentage of re-epithelialization | 100 (0.0)

10. Other Pre Specified Outcome: Achievement of Re-epithelialization - 3 Months
Description: Achievement of re-epithelialization by facial zone and across facial zones after treatment
Time Frame: 3 Months
Population: Data were not collected at 3 months since all subjects had reported 100% re-epithelization prior to 3 months.
Arm/Group | J-Plasma
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Mean Duration for Study Subject to Feel Comfortable in Public After Treatment
Description: Mean duration for study subject to feel comfortable in public after treatment as reported by the subject
Time Frame: Up to 3 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
days | 8.5 (2.5)

12. Other Pre Specified Outcome: Study Subject - Pain/Discomfort Daily 10-point Visual Analog Scale (VAS) Pre-procedure, Post-procedure, and Daily Through the 10 Day Follow-up Visit (10d FUV Visit Window: 9-14 Days)
Description: Daily 10-point Visual Analog Scale (VAS) pain assessments following treatment through the 10 day follow-up visit by diary day with a change from the VAS pain score at baseline. The 10 day follow-up visit window was 9-14 days. Not all participants recorded their VAS score every day on the daily diary; daily diary was collected from each participant at their 10 day follow-up visit (visit window: 9-14 days).
Time Frame: Pre-procedure, post-procedure and Daily through 10 Day Follow-up Visit, approximately 9-14 days
Population: Pain scores on the Visual Analog Scale (VAS) were recorded on a daily diary and analyzed out to the 10 day follow-up visit, with a visit window of 9-14 days. Not all participants recorded a VAS score for each day on the daily diary. Participants' diaries were collected at their 10 day follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
score on a scale
  Pre-procedure 10-point Visual Analog Scale (VAS) | 0.1 (0.4)
  Immediately Post-Procedure 10-point Visual Analog | 4.3 (2.6)
  Day 0 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 54
  Day 0 10-point Visual Analog Scale (VAS) | 3.7 (3.2)
  Day 1 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 54
  Day 1 10-point Visual Analog Scale (VAS) | 2.6 (2.6)
  Day 2 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 52
  Day 2 10-point Visual Analog Scale (VAS) | 2.9 (2.4)
  Day 3 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 53
  Day 3 10-point Visual Analog Scale (VAS) | 2.7 (2.2)
  Day 4 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 53
  Day 4 10-point Visual Analog Scale (VAS) | 3.1 (2.5)
  Day 5 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 52
  Day 5 10-point Visual Analog Scale (VAS) | 3.1 (2.6)
  Day 6 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 52
  Day 6 10-point Visual Analog Scale (VAS) | 2.8 (2.6)
  Day 7 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 51
  Day 7 10-point Visual Analog Scale (VAS) | 2.4 (2.2)
  Day 8 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 52
  Day 8 10-point Visual Analog Scale (VAS) | 2.1 (2.2)
  Day 9 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 50
  Day 9 10-point Visual Analog Scale (VAS) | 1.9 (2.3)
  Day 10 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 42
  Day 10 10-point Visual Analog Scale (VAS) | 1.6 (2.4)
  Day 11 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 26
  Day 11 10-point Visual Analog Scale (VAS) | 1.6 (2.5)
  Day 12 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 17
  Day 12 10-point Visual Analog Scale (VAS) | 1.4 (2.7)
  Day 13 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 12
  Day 13 10-point Visual Analog Scale (VAS) | 1.3 (2.5)
  Day 14 10-point Visual Analog Scale (VAS): number analyzed (Participants) | 6
  Day 14 10-point Visual Analog Scale (VAS) | 1.8 (3.6)

13. Other Pre Specified Outcome: Proportion of Subjects With Correct Identification of 3-month Images
Description: The proportion of subjects (i.e. percentage of treatment responders) with correct identification of 3-month images, in comparison to baseline, as determined by at least 2 out of 3 blinded Independent Photographic Reviewers.
Time Frame: Baseline to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | J-Plasma
Number analyzed (Participants) | 55
Participants | 54

ADVERSE EVENTS:
Time Frame: Through 6 month follow-up visit for all enrolled subjects.
Arm/Group | J-Plasma
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55
Other Adverse Events (participants affected / at risk) | 39/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | J-Plasma (N=55)
Acne (Skin and subcutaneous tissue disorders) | 5 (5)
Hypersensitivity to the treatment (resulting in erythema, swelling, induration, and/or urticaria) (Skin and subcutaneous tissue disorders) | 26 (29)
Itching (Skin and subcutaneous tissue disorders) | 4 (4)
Pain (Skin and subcutaneous tissue disorders) | 3 (3)
Post-inflammatory hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 (8)
Prolonged wound healing (Skin and subcutaneous tissue disorders) | 4 (4)
Sensitivity to topical care (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03286283/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT03286283/SAP_001.pdf